CLINICAL TRIAL: NCT04985916
Title: Clinical Trial to Evaluate ET-01 in Subjects With Lateral Canthal Lines
Brief Title: ET-01 in Subjects With Lateral Canthal Lines, LCL-210
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eirion Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ET-01-LCL-210
Record Dates: First submitted 2021-07-22; First posted 2021-08-02 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Lateral Canthal Lines, LCL; Crow's Feet
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: vehicle controlled, parallel group
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vehicle (Placebo Comparator): Vehicle, topical liniment, administered once at baseline
  Interventions: Biological: Vehicle
- ET-01, Dose 1 (Experimental): Dose 1 of botulinum toxin, Type A, topical liniment, administered once at baseline. 250µm microneedle length
  Interventions: Biological: botulinum toxin, Type A
- ET-01, Dose 2 (Experimental): Dose 2 of botulinum toxin, Type A, topical liniment, administered once at baseline. 250µm microneedle length
  Interventions: Biological: botulinum toxin, Type A

INTERVENTIONS:
Biological: Vehicle — topical liniment without investigational product
  Other Names: ET-01 Vehicle
  Arms: Vehicle
Biological: botulinum toxin, Type A — ET-01 topical liniment
  Other Names: ET-01
  Arms: ET-01, Dose 1; ET-01, Dose 2

SUMMARY:
This study tests an investigational drug formulation called ET-01, botulinum toxin, Type A, topical, in lateral canthal lines (LCL).

DETAILED DESCRIPTION:
This product is being tested for its ability to reduce lateral canthal lines (LCL), also known as Crow's Feet.

ELIGIBILITY:
Inclusion Criteria:

* able to understand and give written informed consent
* 25 - 65 years of age
* willing to have facial pictures/videos taken per protocol
* mild or less Crow's Feet wrinkles (IGA 0-2) "at rest"
* moderate to severe Crow's Feet (IGA 3-4) "on contraction"
* ability to correctly grade a series of Crow's Feet pictures
* moderate to severe Crow's Feet (SSA 3-4) "on contraction"
* have adequate vision without the use of eyeglasses to assess facial wrinkles in a mirror (contact lenses are OK)
* willingness to refrain from the use of facial fillers, retinoids, botulinum toxins, laser treatments, or any product affecting skin remodeling or that might cause an active dermal response during the course of the study
* female subjects of childbearing potential must have a negative urine pregnancy test and be non-lactating at the Baseline visit
* female subjects of childbearing potential must utilize one of the following methods of birth control throughout the study: intra-uterine device (IUD), diaphragm, a condom, a spermicidal gel or foam, oral contraceptives (provided subject has been utilizing this method for at least 3 months prior to Baseline and has not changed the brand within this period), or patch, injectable, implantable, or vaginal ring contraceptives. Subjects may also participate if they are surgically sterilized (tubal sterilization or hysterectomy) or are in menopause.
* subjects should be in good general health as determined by the Investigator and free of any disease that may interfere with study evaluations or the Investigational Product.

Exclusion Criteria:

* history of adverse reactions to any prior botulinum toxin treatments
* history of vaccination with botulinum toxin
* history of non-response to any prior botulinum toxin treatments
* any botulinum toxin treatment anywhere in the prior 6 months
* history of participation in ET-01-LCL-210 in previous Cohorts 1 or 2 at any time in the past
* history of periocular surgery, brow lift or related procedures
* soft tissue augmentation or any procedures affecting the lateral canthal region in the prior 12 months
* dermabrasion or laser treatment in the periocular region in the last 6 months
* topical prescription-strength retinoids in the prior 3 months to the treatment area
* application of any topical prescription medication to the treatment area within 14 days prior to treatment
* subjects on clinically significant, concomitant drug therapy (See Section 5.3 below).).
* present or history of neuromuscular disease, eyelid ptosis, muscle weakness or paralysis
* present or history of "dry eye"
* hemophilia, hemorrhagic disorder, hemostatic dysfunction or other blood clotting disorders
* use of systemic aminoglycosides in the week prior to treatment application
* participation in another investigational drug trial or receiving any investigational treatment(s) within 30 days of Baseline
* alcohol or drug abuse within the past 3 years
* psychiatric disease interfering with the subject's ability to give informed consent
* refusal or inability to comply with the requirements of the protocol for any reason

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
IGA (Investigators Global Assessment) | Week 4
  Investigators Global Assessment. Crow's Feet Wrinkle Scale where severity is scored between 0-4 (0=absent; 4=severe).

SECONDARY OUTCOMES:
IGA (Investigators Global Assessment) | Week 2, 4, 8,12, and 18
  Investigators Global Assessment. Crow's Feet Wrinkle Scale where severity is scored between 0-4 (0=absent; 4=severe).
SSA (Subject Self-Assessment) | Week 2, 4, 8,12, and 18
  Subject Self-Assessment. Crow's Feet Wrinkle Scale where severity is scored between 0-4 (0=absent; 4=severe).

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Eirion Research Site, Scottsdale, Arizona
  - Eirion Research Site, San Diego, California
  - Eirion Research Site, Aventura, Florida
  - Eirion Research Site, Boca Raton, Florida
  - Eirion Research Site, Miami, Florida
  - Eirion Research Site, West Palm Beach, Florida
  - Eirion Research Site, Chicago, Illinois
  - Eirion Research Site, Louisville, Kentucky
  - Eirion Research Site, New Orleans, Louisiana
  - Eirion Research Site, Glenn Dale, Maryland
  - Eirion Research Site, Clinton Township, Michigan
  - Eirion Research Site, New Brighton, Minnesota
  - Eirion Research Site, New York, New York
  - Eirion Research Site, Exton, Pennsylvania
  - Eirion Research Site, Newtown Square, Pennsylvania
  - Eirion Research Site, Greenville, South Carolina
  - Eirion Research Site, Houston, Texas
  - Eirion Research Site, Plano, Texas
  - Eirion Research Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No